CLINICAL TRIAL: NCT05909410
Title: Perception About Benefits and Risks Related to Combined Hormonal Contraceptives Use in Patients With Lynch Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, principal investigator, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: HORMONES-LYNCH
Record Dates: First submitted 2023-05-26; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Lynch Syndrome; Contraception
Keywords: Lynch syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Lynch syndrome: Certain genetic diagnosis o fLynch syndrome
  Interventions: Other: Survey investigating the CHC use and patients' perception about the relationship between CHC and cancer, diseases and symptoms
- Healthy patients of reproductive age
  Interventions: Other: Survey investigating the CHC use and patients' perception about the relationship between CHC and cancer, diseases and symptoms

INTERVENTIONS:
Other: Survey investigating the CHC use and patients' perception about the relationship between CHC and cancer, diseases and symptoms — This survey investigated the CHC use (type and timing of administration) and patients' perception about the relationship between CHC and cancer, diseases and symptoms

SUMMARY:
Combined hormonal contraceptives (CHCs), according to the opinion by The Manchester International Consensus Group, should be considered for women wishing contraception because also positively impact endometrial cancer and ovarian cancer risk. The awareness of the effects of hormonal therapies in women at high risk of developing endometrial cancer, colorectal, breast, or ovarian cancer, such as those affected by Lynch syndrome (LS), is currently limited, with few published studies addressing these populations. Making informed decisions about CHC use in this context necessitates careful consideration of individual cancer risk and the potential benefits and risks associated with CHC use. Accurate information regarding the oncological risks associated with CHC use is essential for facilitating shared decision-making between women and their healthcare providers in this patient population.

This prospective study aims to evaluate the knowledge, attitudes, and beliefs of women with LS concerning CHCs and their potential effects on specific disease development and cancer risk, comparing them to the general population. By considering psychosocial factors and individual perceptions of cancer risk, this study seeks to contribute to informed decision-making, personalized counseling, and improved strategies for gynecologic cancer risk management in women with LS.

ELIGIBILITY:
Inclusion Criteria:

* patients with certain genetic diagnosis of Lynch syndrome and patients of reproductive age undergoing routinely gynecological visit

Exclusion Criteria:

* for both groups, a prior history of oncological diseases and a personal history of endometrial cancer, colorectal cancer, ovarian cancer, or breast cancer.
* for patients with Lynch syndrome, individuals who had undergone previous risk-reducing prophylactic surgical approaches such as (risk-reducing) colectomy, hysterectomy, early salpingectomy, and delayed oophorectomy, and risk-reducing salpingo-oophorectomy

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Study Population: Patients with certain genetic diagnosis of Lynch syndrome and of reproductive age undergoing routinely gynecological visit
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients using currently CHCs | Through study completion, an average of 1 month
  Evaluation of the number (%) of patients using currently CHCs
Number of patients having used CHCs | Through study completion, an average of 1 month
  Evaluation of the number (%) of patients having used CHCs in the past
Perception about the impact of CHCs on favoring/contrasting specific cancer onset | Through study completion, an average of 1 month
  By using a Likert scale (from -5 to +5)
Perception about the impact of CHCs on favoring/contrasting specific chronic disease onset | Through study completion, an average of 1 month
  By using a Likert scale (from -5 to +5)
Perception about the impact of CHCs on favoring/contrasting specific symptoms onset | Through study completion, an average of 1 month
  By using a Likert scale (from -5 to +5)

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ferrero, Principal Investigator — Piazza della Vittoria 14
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grandi G, Monari F, Boggio Sola V, Cortesi L, Toss A, Del Savio MC, Melotti C, Centurioni MG, Gustavino C, Varesco L, Facchinetti F, Barra F. BRCA mutation carriers' perception about benefits and risks associated with combined hormonal contraceptives use. Eur J Contracept Reprod Health Care. 2022 Dec;27(6):439-444. doi: 10.1080/13625187.2022.2107199. Epub 2022 Aug 10. PMID 35946412
- [Background] Grandi G, Boggio Sola V, Cortesi L, Toss A, Giuliani GA, Del Savio MC, Facchinetti F. BRCA mutation carriers' perceptions on postmenopausal hormone therapy: An Italian study. Psychooncology. 2021 Oct;30(10):1711-1719. doi: 10.1002/pon.5714. Epub 2021 May 28. PMID 34002428
- [Background] Grandi G, Del Savio MC, Boggio Sola V, Monari F, Melotti C, Facchinetti F. Attitudes of women towards products containing hormones (hormonal contraceptives or hormone therapy): what changes from pre to postmenopause? Ann Med. 2021 Dec;53(1):908-915. doi: 10.1080/07853890.2021.1938662. PMID 34124968